CLINICAL TRIAL: NCT04799184
Title: Pharmacokinetics and Pharmacodynamics for Levobupivacaine with and Without Epinephrine After Ultrasound Guided Erector Spinae Plane Block
Brief Title: PK/PD Levobupivacaine with and Without Epinephrine After Ultrasound Guided ESP Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170627010
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Anesthetics Complications; Anesthetic Toxicity; Bupivacaine Overdose; Nerve Block; Surgery
Keywords: ESP; Perioperative Care; Bupivacaine Overdose; VATS surgery
MeSH Terms: interventions — Levobupivacaine; Epinephrine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups, this will be done through a table of computer-generated random numbers.
  Group I will receive ESP block with vasoconstrictor and Group II will receive ESP block without vasoconstrictor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I Epi (Experimental): The ESP will be performed under ultrasound vision at T5 level, with the patient seated.
  Once the ultrasound image is achieved, a 100 mm, 20 G Stimuplex needle will be punctured and a solution of levobupivacaine 0.25% with epinephrine 5 ug/ml completing a volume of 20 ml.
  Interventions: Drug: Levobupivacaine 0.25% with epinephrine 5 ug/ml
- Group II no Epi (Active Comparator): The ESP will be performed under ultrasound vision at T5 level, with the patient seated.
  Once the ultrasound image is achieved, a 100 mm, 20 G Stimuplex needle will be punctured and a solution of levobupivacaine 0.25% without epinephrine completing a volume of 20 ml.
  Interventions: Drug: Levobupivacaine 0.25% without epinephrine 5 ug/ml

INTERVENTIONS:
Drug: Levobupivacaine 0.25% with epinephrine 5 ug/ml — The block will be performed under ultrasound vision at T5 level, with the patient seated.
  Once the ultrasound image is achieved, a 100 mm, 20 G Stimuplex needle will be punctured and a solution of levobupivacaine 0.25% with epinephrine 5 ug / ml until completing a volume of 20 ml in fractional form.
  Other Names: ESP; Bupivacaine
  Arms: Group I Epi
Drug: Levobupivacaine 0.25% without epinephrine 5 ug/ml — The block will be performed under ultrasound vision at T5 level, with the patient seated.
  Once the ultrasound image is achieved, a 100 mm, 20 G Stimuplex needle will be punctured and a solution of levobupivacaine 0.25% without epinephrine 5 ug / ml until completing a volume of 20 ml in fractional form.
  Other Names: ESP; Bupivacaine
  Arms: Group II no Epi

SUMMARY:
Currently there is no standardized management or single technique to manage postoperative pain after Video-assisted thoracic surgery (VATS), there are many options available ranging from intravenous opioids, morphine or fentanyl Patient-controlled analgesia (PCA), peripheral nerve blocks, intercostals, paravertebral and epidural blocks. Erector Spinal Block (ESP), this blocks the ventral and dorsal branch of the unilateral thoracic roots. It corresponds to an interfacial block that produces an extensive multidermatomal sensitive block with a single puncture, covering the anterior, lateral and posterior aspect of the thorax. One of its main advantages would be safety, possible less damage to nerves and pneumothorax, as well as the simplicity of execution of this block. What has positioned it as another analgesic alternative in this type of surgery.

The pharmacokinetic profile that local anesthetics would have when injected into this interfacial compartment has not yet been described, and what the real impact of the use of vasoconstrictor will be in terms of plasma levels and duration of the block.

Our objective is to compare the plasma levels of levobupivacaine achieved after performing an ESP Block with or without epinephrine.

DETAILED DESCRIPTION:
Video-assisted thoracic surgery (VATS) is one of the most common procedures performed in thoracic surgery, mainly because it has made it possible to solve many pathologies that previously required a thoracotomy with all the complications that that meant. VATS has been shown to be beneficial for patients, for many reasons such as lower mortality, better postoperative lung function, and shorter stay during hospitalization.

Less invasive procedures such as VATS, where the surgical incision is small and avoids costal resection, produces less postoperative pain when compared to a thoracotomy, this has been objectified by numerous studies that have found lower scores on the numerical verbal scale (NVE) and fewer requirements for pain relievers. Despite the fact that VATS produces less acute postoperative pain (VNS 4-5 on the first postoperative day in VATS vs VNS 6 in thoracotomies), the incidence of chronic postoperative pain ranges from 20 to 47%, which is comparable to thoracotomy, mainly due to damage to the intercostal nerves and inadequate analgesia.

It has been seen that one of the factors associated with the appearance of chronic pain after chest surgery is severe acute pain in the first three postoperative days. Acute pain in VATS is caused by surgical trauma to muscular and bone structures of the thorax, achieving good analgesia is important to maintain adequate respiratory function and avoid complications such as atelectasis, hypoxemia and possible pneumonia.

Currently, there is no standardized management or single technique to manage postoperative pain after VATS, there are many options available ranging from intravenous opioids, morphine or fentanyl Patient-controlled analgesia, peripheral nerve blocks, intercostals, paravertebral and epidural blocks. Each of them with advantages and disadvantages, but without being able to demonstrate a clear superiority between them, both the paravertebral and epidural blocks are the ones that accumulate the most reports in the literature regarding the management of postoperative pain, but at the same time they are not exempt from complications such as technical failure, hypotension and difficulty of the procedure. In addition to documenting a low use of thoracic epidurals in VATS.

At the end of 2016, the description of the Erector Spinal Block (ESP) by Forero was published, it blocks the ventral and dorsal branch of the unilateral thoracic roots. It corresponds to an interfacial block that produces an extensive multidermatomal sensitive block with a single puncture, covering the anterior, lateral and posterior aspect of the thorax. One of its main advantages would be safety, possible less nerve damage and pneumothorax, as well as the simplicity of execution of this block. What has positioned it as another analgesic alternative in this type of surgery.

In ESP, the pharmacokinetic (PK) profile that local anesthetics would have when injected into this interfacial compartment has not yet been described, and what will be the real impact of the use of vasoconstrictor in terms of plasma levels and duration of the block.

Considering the above, it is important to know the pharmacodynamics of levobupivacaine after performing an ESP block with ultrasonography in order to know the risks of toxicity from local anesthetics as well as to clinically characterize this block in patients who will undergo VATS.

The first objective of this study is to compare the plasma levels of levobupivacaine achieved after performing an ESP Block with or without epinephrine. As secondary objectives, it is proposed to characterize the block in terms of duration, pain, opioid requirements in the first 24 hours and adverse events, in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Indication of VATS
* ASA I-II
* Body mass index (BMI) 20-34 kg / m2

Exclusion Criteria:

* Patients with conversion to thoracotomy
* History of chronic pain
* Drug abuse
* Psychiatric illness
* Allergic to some of the drugs used in the study
* Chronic analgesic users
* History of peripheral neuropathy
* Who refuse the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Plasma levels of levobupivacaine | 5, 10, 20, 30, 60, 90 minutes post block.
  Levobupivacaine plasma levels will be measured using High-performance liquid chromatography.
Changes in plasma levels levobupivacaine of the group I v/s group II | 5, 10, 20, 30, 60, 90 minutes post block.
  To assess the changes in plasma levels of the group I with epinephrine versus the group II without epinephrine.
Sensitive skin extension | 15 minutes post-block
  Determine the sensitive skin extension of ESP after its performance using pinprick and temperature discrimination using an alcohol swab.

SECONDARY OUTCOMES:
Pain measured | Every 15 minutes per 2 hours in the PACU and 12 hrs, 24 hrs, 48 hrs during hospitalization
  Pain measured by Verbal Numerical Scale (VNS) 0 to 10. 0 = no pain. 10 = worse pain.
Heart Rate | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  Heart rate (bpm)
Hemodynamics | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  Invasive arterial pressure (mmHg)
Pulse oximetry | Every 5 min. Since entering operating room up to end of anesthesia and leaving to recovery room. In average 2 hrs.
  % oximetry saturation
Consumption of morphine or its equivalents | During the first 48 hours including intraoperative and postoperative
  Consumption of morphine or its equivalents (mg/kg/hr)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Araneda, MD, Principal Investigator — Clinician
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Procedure performance of ESP in terms of duration and user satisfaction
Supporting Information: Study Protocol
Time Frame: After the paper publication
Access Criteria: Researchers and clinicians related to the analgesic management of patients, upon formal request via e-mail to the research director.

REFERENCES:
- [Background] Corvetto MA, Echevarria GC, De La Fuente N, Mosqueira L, Solari S, Altermatt FR. Comparison of plasma concentrations of levobupivacaine with and without epinephrine for transversus abdominis plane block. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):633-7. doi: 10.1097/AAP.0b013e31826c330a. PMID 23038415
- [Derived] Araneda A, De la Cuadra JC, Corvetto M, Balde D, Fuente R, Ibacache M, Contreras V, Solari S, Cortinez I. Pharmacokinetic modelling and simulation for prolonged infusion of levobupivacaine with or without epinephrine in transversus abdominis plane and erector spinae plane blocks: a randomised controlled trial and analysis of pooled data. Br J Anaesth. 2025 Oct;135(4):1051-1058. doi: 10.1016/j.bja.2025.05.047. Epub 2025 Jul 9. PMID 40640046